CLINICAL TRIAL: NCT06389487
Title: A Phase 3b, Open-label Study to Evaluate the Non-inferiority of the Immune Response and to Evaluate the Safety of the RSVPreF3 OA Investigational Vaccine in Adults 18-49 Years of Age at Increased Risk for Respiratory Syncytial Virus Disease, Compared to Older Adults >=60 Years of Age
Brief Title: A Study on the Immune Response and Safety of Vaccine Against Respiratory Syncytial Virus (RSV) Given to Adults 18 to 49 Years of Age at Increased Risk for Respiratory Syncytial Virus Disease, Compared to Older Adults 60 Years of Age and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 222253; 2023-510190-34-00 (Other: EU CTR Number)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); Immunogenicity; Safety; Non-inferiority; Humoral immune response; At increased risk (AIR); Older Adults
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: RSV-A-AIR Group (Experimental): Adult (A) participants, 18-49 YOA, at increased risk (AIR) for RSV disease, received a single dose of RSVPreF3 OA investigational vaccine at Day 1. Participants in this group were considered for all study analyses, as per protocol.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Part A: RSV-OA Group (Active Comparator): Older adults (OA) participants, ≥60 YOA, received a single dose of RSVPreF3 OA investigational vaccine at Day 1.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Part B: RSV-A-AIR Group (Experimental): Adult participants, 18-49 YOA, AIR for RSV disease, received a single dose of RSVPreF3 OA investigational vaccine at Day 1. Participants in this group were considered only for Participant flow, Baseline Characteristics and all safety analyses, as per protocol.
  Interventions: Biological: RSVPreF3 OA investigational vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — 1 dose of RSVPreF3 OA investigational vaccine is administered intramuscularly on Day 1.

SUMMARY:
The aim of this study is to demonstrate the immune response and to evaluate the safety of the RSVPreF3 OA investigational vaccine in non-immunocompromised adults 18-49 years of age (YOA), who are at increased risk (AIR) for RSV disease, compared to older adults (OA) 60 YOA and above.

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or participant's parent(s)/ Legally acceptable representative (LAR) who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, attend study site visits, ability to access and utilize a phone or other electronic communications).
* Written or witnessed informed consent obtained from the participant/participant's parent(s)/LAR(s) (participant must be able to understand the informed consent) prior to performance of any study-specific procedure.

Written informed assent obtained from the participant (participant must be able to understand the informed assent) if he/she is less than the legal age prior to performance of any study-specific procedure.

Specific inclusion criteria for all participants in Cohort 1 and Cohort 3 (RSV-A-AIR Group) • A male or female participant 18-49 YOA at the time of the study intervention administration.

* Participants should be diagnosed with at least 1 of the following medical conditions if considered medically stable by the investigator:

  * Chronic cardiopulmonary disease resulting in activity restricting symptoms or use of long term medication:

    o Chronic obstructive pulmonary disease (COPD)

    o Asthma

    o Cystic fibrosis

    o Other chronic respiratory diseases: lung fibrosis, restrictive lung disease, interstitial lung disease, emphysema or bronchiectasis

    o Chronic heart failure:

    o Pre-existing Coronary Artery Disease (CAD) (CAD not otherwise specified)
    * Cardiac arrhythmia
  * Diabetes mellitus: types 1 or 2 with active treatment for the past 6 months
  * Other diseases at increased risk for RSV disease:

    * Chronic kidney disease
    * Chronic moderate to severe liver disease
    * Neurologic or neuromuscular conditions
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as premenarche, hysterectomy, bilateral oophorectomy, bilateral salpingectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception from 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study prior to intervention administration, and
  * has agreed to continue adequate contraception for at least 1 month after completion of the study intervention administration.

Specific inclusion criteria for all participants in Cohort 2 (RSV-OA Group):

• A male or female participant >=60 YOA at the time of the study intervention administration.

Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease are allowed to participate in this study if considered medically stable by the investigator.

• Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., current malignancy, human immunodeficiency virus) or immunosuppressive/cytotoxic therapy (e.g., medication used during cancer chemotherapy, organ transplantation, or to treat autoimmune disorders), based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol (e.g., completion of the diary cards, attend study site visits). Study participants may decide to assign a caregiver to help them complete the study procedures.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease).
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study intervention during the period beginning 30 days before the dose of study intervention (Day -29 to Day 1), or planned use during the study period (up to Visit 3, Month 6).
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of study intervention administration, with the exception of inactivated, subunit and split influenza vaccines or COVID-19 vaccines which can be administered up to 14 days before or from 14 days after the study intervention administration.
* Previous vaccination with any RSV vaccine, including investigational RSV vaccines.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or administration of long-acting immune-modifying treatments or planned administration at any time up to the End-of-study (EOS).

  * Up to 3 months prior to the study intervention administration:

    * For corticosteroids, this will mean prednisone >=20 mg/day, or equivalent. Inhaled, topical and intra-articular steroids are allowed
    * Administration of immunoglobulins and/or any blood products or plasma derivatives
  * Up to 6 months prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy (e.g., Tumor Necrosis Factor (TNF)-inhibitors), monoclonal antibodies, antitumoral medication.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or invasive medical device).

Other exclusions:

Other exclusions for all participants:

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study period that will prohibit participating in the study until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.

Other exclusions for Cohort 1 and Cohort 3:

* Pregnant or lactating female participant.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 1 month after study intervention administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1459 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2025-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (16):
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, North Hollywood, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Wenatchee, Washington
- Australia (6):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Fortitude Valley, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, St Albans, Victoria
- Canada (10):
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, London-Ontario, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (7):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Wallerfing
  - GSK Investigational Site, Witten
  - GSK Investigational Site, Würzburg
- Japan (3):
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- South Africa (3):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Reiger Park

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1459 participants were enrolled, out of which 1458 were included in the Exposed set and started the study.
Groups:
- Part A: RSV-A-AIR Group: Adult (A) participants, 18-49 years of age (YOA), at increased risk (AIR) for respiratory syncytial virus (RSV) disease, received a single dose of RSVPreF3 OA investigational vaccine at Day 1. Participants in this group were considered for all study analyses, as per protocol.
- Part A: RSV-OA Group: Older adults (OA) participants, greater than or equal to (≥) 60 YOA, received a single dose of RSVPreF3 OA investigational vaccine at Day 1.
Period: Overall Study
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Started | 426 | 429 | 603
Completed | 414 | 422 | 586
Not Completed | 12 | 7 | 17
Not completed — Lost to Follow-up | 9 | 5 | 13
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A: RSV-A-AIR Group: Adult participants, 18-49 years of age (YOA), at increased risk (AIR) for respiratory syncytial virus (RSV) disease, received a single dose of RSVPreF3 OA investigational vaccine at Day 1. Participants in this group were considered for all study analyses, as per protocol.
- Total: Total of all reporting groups
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group | Total
Number analyzed (Participants) | 426 | 429 | 603 | 1458
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 38.9 (7.8) | 68.6 (5.7) | 38.1 (8.7) | 47.3 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 220 | 347 | 814
  Male | 179 | 209 | 256 | 644
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 0 | 11 | 19
  Asian | 60 | 50 | 64 | 174
  Balck or African American | 77 | 54 | 181 | 312
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 11 | 11
  White | 255 | 302 | 274 | 831
  Not reported | 3 | 1 | 0 | 4
  Unknown | 4 | 0 | 3 | 7
  Multiple Race Categories | 19 | 22 | 59 | 100

OUTCOME MEASURES:

1. Primary Outcome: Part A: RSV-A Neutralizing Titers Expressed as Group Geometric Mean Titers (GMTs)
Description: RSV-A neutralizing titers are given as group GMTs and are expressed as Estimated dilution 60 (ED60)
Time Frame: At Day 31
Population: Analysis was performed on the per protocol set (PPS) which included all eligible participants who received the study intervention as per protocol, had RSV-A immunogenicity results pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on age and medical condition including participants with data available at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 393 | 417
Titer | 11910.1 [10927.3 to 12981.4] | 8593.6 [7904.3 to 9343.0]
Statistical Analysis 1: Comparison: Part A: RSV-A-AIR Group vs Part A: RSV-OA Group; To demonstrate the non-inferiority of the humoral immune response in participants aged 18-49 YOA at increased risk for RSV disease (Part A:RSV-A-AIR Group) compared to older adults aged ≥60 YOA (Part A:RSV-OA Group) for the RSV-A strain after RSVPreF3 OA investigational vaccine administration; Test type: Non-Inferiority — Non-Inferiority (NI) was to be demonstrated if the upper limit of the 95% confidence interval (CI) of the group GMT ratio between Part A:RSV-OA Group over Part A:RSV-A-AIR Group at 1 month post RSVPreF3 OA vaccine administration was less than or equal to (≤) 1.5; GMT Ratio = 0.72, 95% CI 2-sided [0.64 to 0.81] — The comparison is done using the group ratio of adjusted GMT (Part A:RSV-OA/ Part A:RSV-A-AIR) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate

2. Primary Outcome: Part A: Percentage of Participants With Seroresponse Rate (SRR) in RSV-A Neutralizing Titers
Description: SRR is defined as the percentage of participants having a fold increase in neutralizing titers (1 month post-study intervention administration over pre-study intervention administration) ≥4. RSV-A neutralizing titers are expressed as ED60.
Time Frame: Day 31 compared with baseline (Day 1)
Population: Analysis was performed on the PPS which included all eligible participants who received the study intervention as per protocol, had RSV-A immunogenicity results pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on age and medical condition including participants with data available at specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 342 | 324
Percentage of participants | 87.0 [83.3 to 90.2] | 77.7 [73.4 to 81.6]
Statistical Analysis 1: Comparison: Part A: RSV-A-AIR Group vs Part A: RSV-OA Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 95% CI of the group SRR difference between Part A:RSV-OA Group and Part A:RSV-A-AIR Group at 1 month post RSVPreF3 OA vaccine administration was ≤10%; Difference in percentage = -9.33, 95% CI 2-sided [-14.55 to -4.10] — The comparison is done using the difference of SRR (Part A:RSV-OA - Part A:RSV-A-AIR)

3. Primary Outcome: Part A: RSV-B Neutralizing Titers Expressed as Group GMTs
Description: RSV-B neutralizing titers are given as group GMTs and are expressed as ED60.
Time Frame: At Day 31
Population: Analysis was performed on the PPS which included all eligible participants who received the study intervention as per protocol, had RSV-B immunogenicity results pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on age and medical condition including participants with data available at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 392 | 417
Titer | 12496.4 [11482.4 to 13599.9] | 9089.7 [8373.7 to 9866.9]
Statistical Analysis 1: Comparison: Part A: RSV-A-AIR Group vs Part A: RSV-OA Group; To demonstrate the non-inferiority of the humoral immune response in participants aged 18-49 YOA at increased risk for RSV disease (Part A:RSV-A-AIR Group) compared to older adults aged ≥60 YOA (Part A:RSV-OA Group) for the RSV-B strain after RSVPreF3 OA investigational vaccine administration; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 95% CI of the group GMT ratio between Part A:RSV-OA Group over Part A:RSV-A-AIR Group at 1 month post RSVPreF3 OA vaccine administration was ≤1.5; GMT Ratio = 0.73, 95% CI 2-sided [0.65 to 0.82] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Part A: Percentage of Participants With SRR in RSV-B Neutralizing Titers
Description: SRR is defined as the percentage of participants having a fold increase in neutralizing titers (1-month post-study intervention administration over pre-study intervention administration) ≥ 4. RSV-B neutralizing titers are expressed as ED60.
Time Frame: Day 31 compared with baseline (Day 1)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 342 | 322
Percentage of participants | 87.2 [83.5 to 90.4] | 77.2 [72.9 to 81.2]
Statistical Analysis 1: Comparison: Part A: RSV-A-AIR Group vs Part A: RSV-OA Group; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -10.03, 95% CI 2-sided [-15.26 to -4.80] — The comparison is done using the difference of SRR (Part A:RSV-OA - Part A:RSV-A-AIR)

5. Secondary Outcome: Part A and B: Number of Participants Reporting Any Solicited Administration Site Events
Description: Assessed solicited administration site events were pain, redness (erythema) and swelling at administration site. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Day 1 (post dose) to Day 4
Population: Analysis was performed on the Exposed Set, which included all participants who received the study intervention. Analysis per group is based on age and medical condition. Only those participants with solicited administration site events were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Number analyzed (Participants) | 425 | 428 | 601
Participants
  Pain | 358 | 246 | 422
  Redness | 36 | 23 | 52
  Swelling | 25 | 19 | 47

6. Secondary Outcome: Part A and B: Number of Participants Reporting Any Solicited Systemic Events
Description: Assessed solicited systemic events were fever (pyrexia), headache, myalgia (muscle pain), arthralgia (joint pain) and fatigue (tiredness). Fever was defined as temperature ≥38.0 degrees Celsius (°C), regardless of the location of measurement. The route for measuring temperature could be oral or axillary. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Day 1 (post dose) to Day 4
Population: Exposed Set. Only those participants with solicited systemic events were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Number analyzed (Participants) | 425 | 428 | 602
Participants
  Fever | 25 | 11 | 26
  Headache | 198 | 78 | 250
  Myalgia | 284 | 169 | 331
  Arthralgia | 124 | 78 | 167
  Fatigue | 275 | 148 | 337

7. Secondary Outcome: Part A and B: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AE wass an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs included both serious and non-serious AEs.
Time Frame: Day 1 (post dose) to Day 30
Population: Exposed Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Number analyzed (Participants) | 426 | 429 | 603
Participants | 72 | 76 | 118

8. Secondary Outcome: Part A and B: Number of Participants Reporting Any Serious Adverse Events (SAEs), Related SAEs and Fatal SAEs
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is considered or defined as an important medical event, or abnormal pregnancy outcomes. Any SAE = occurrence of the SAE regardless of the intensity grade or relation to study vaccination. Related SAE = SAE assessed by the investigator as related to the study vaccination. Fatal SAE = occurrence of a fatal SAE regardless of relation to study vaccination.
Time Frame: Throughout the study period (Day 1 to Month 6)
Population: Exposed Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Number analyzed (Participants) | 426 | 429 | 603
Participants
  Any SAEs | 4 | 13 | 10
  Related SAEs | 0 | 0 | 0
  Fatal SAEs | 0 | 0 | 0

9. Secondary Outcome: Part A and B: Number of Participants Reporting Any Adverse Events of Special Interest (AESIs)
Description: AESIs assessed were potential immune-mediated diseases (pIMDs) and atrial fibrillation (AF). pIMDs were a subset of AESIs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. AEs of AF were considered as AESI.
Time Frame: Throughout the study period (Day 1 to Month 6)
Population: Exposed Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
Number analyzed (Participants) | 426 | 429 | 603
Participants | 1 | 2 | 2

10. Secondary Outcome: Part A: RSV-A Neutralizing Titers Expressed as GMTs
Description: RSV-A neutralizing titers are given as GMTs and are expressed as ED60.
Time Frame: At Day 1 (pre-dose), at Month 1 and Month 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 419 | 425
Titer
  Day 1 | 892.6 [821.5 to 969.9] | 913.8 [837.2 to 997.4]
  Month 1: number analyzed (Participants) | 393 | 417
  Month 1 | 11853.4 [10875.3 to 12919.5] | 8632.4 [7858.3 to 9482.6]
  Month 6: number analyzed (Participants) | 393 | 406
  Month 6 | 4439.8 [4042.1 to 4876.7] | 3917.7 [3553.0 to 4319.7]

11. Secondary Outcome: Part A: RSV-B Neutralizing Titers Expressed as GMTs
Description: RSV-B neutralizing titers are given as GMTs and are expressed as ED60.
Time Frame: At Day 1 (pre-dose), at Month 1 and Month 6
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group
Number analyzed (Participants) | 418 | 425
Titer
  Day 1 | 988.1 [905.9 to 1077.8] | 1045.1 [953.7 to 1145.2]
  Month 1: number analyzed (Participants) | 393 | 417
  Month 1 | 12337.6 [11334.3 to 13429.7] | 9178.5 [8367.7 to 10067.8]
  Month 6: number analyzed (Participants) | 393 | 406
  Month 6 | 4335.6 [3941.7 to 4769.0] | 4355.0 [3971.4 to 4775.7]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 (day of vaccination) up to Day 4 post-dose. Unsolicited AEs were collected from Day 1 up to Day 30 post-dose. All-cause mortality, SAEs, related SAEs, fatal SAEs and AESIs (including pIMDs and AF) were collected from Day 1 up to study end (Month 6)
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Part A: RSV-A-AIR Group | Part A: RSV-OA Group | Part B: RSV-A-AIR Group
All-Cause Mortality (participants affected / at risk) | 0/426 | 0/429 | 0/603
Serious Adverse Events (participants affected / at risk) | 4/426 | 13/429 | 10/603
Other Adverse Events (participants affected / at risk) | 386/426 | 310/429 | 483/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: RSV-A-AIR Group (N=426) | Part A: RSV-OA Group (N=429) | Part B: RSV-A-AIR Group (N=603)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of asthma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vulval cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: RSV-A-AIR Group (N=426) | Part A: RSV-OA Group (N=429) | Part B: RSV-A-AIR Group (N=603)
Injection site pain (General disorders) | 358 (364) | 246 (247) | 422 (425)
Fatigue (General disorders) | 275 (284) | 148 (151) | 338 (352)
Injection site erythema (General disorders) | 37 (39) | 23 (23) | 52 (53)
Injection site swelling (General disorders) | 25 (26) | 19 (19) | 47 (47)
Pyrexia (General disorders) | 26 (26) | 12 (12) | 29 (30)
Chills (General disorders) | 5 (5) | 2 (2) | 13 (13)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 7 (7)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 3 (3)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site macule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site plaque (General disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 284 (290) | 169 (170) | 331 (338)
Arthralgia (Musculoskeletal and connective tissue disorders) | 126 (128) | 81 (83) | 167 (171)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 198 (200) | 78 (79) | 250 (258)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain fog (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7) | 10 (10)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 6 (6)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 6 (6)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (14) | 2 (2) | 12 (12)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Auditory disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Metabolic dysfunction-associated liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT06389487/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT06389487/SAP_001.pdf